CLINICAL TRIAL: NCT01076634
Title: A Trial Investigating the Pharmacodynamic Properties of NN1250 in Subjects With Type 1 Diabetes
Brief Title: Comparison of Two NN1250 Formulations in Subjects With Type 1 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NN1250-3678; 2009-014555-68 (EudraCT Number); U1111-1112-7714 (Other: WHO)
Record Dates: First submitted 2010-02-24; First posted 2010-02-26 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — insulin degludec

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- IDeg 100 U/mL (Experimental)
  Interventions: Drug: insulin degludec
- IDeg 200 U/mL (Experimental)
  Interventions: Drug: insulin degludec

INTERVENTIONS:
Drug: insulin degludec — 0.4 U/kg body weight. Injected subcutaneously (under the skin) once daily for 8 days.
  Arms: IDeg 100 U/mL
Drug: insulin degludec — 0.4 U/kg body weight. Injected subcutaneously (under the skin) once daily for 8 days.
  Arms: IDeg 200 U/mL

SUMMARY:
This trial is conducted in Europe. The aim of the trial is to investigate the pharmacodynamic properties (effect) by comparing two NN1250 (insulin degludec, IDeg) formulations in subjects with type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes mellitus (as diagnosed clinically) for at least 12 months
* Body mass index 18.0-28.0 kg/m^2 (both inclusive)

Exclusion Criteria:

* Subject who has donated any blood or plasma in the past month or more than 500 mL within 3 months prior to screening
* Smoker (defined as a subject who is smoking more than 5 cigarettes or the equivalent per day)
* Not able or willing to refrain from smoking and use of nicotine gum or transdermal nicotine patches during the inpatient period

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2010-02; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Area under the glucose infusion rate curve during one dosing interval at steady-date" | After 8 days of treatment

SECONDARY OUTCOMES:
Area under the serum Insulin Degludec concentration-time curve | During one dosing interval at steady state
Area under the serum Insulin Degludec concentration-time curve | From 0 to 24 hours after single dose

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Graz, Austria

REFERENCES:
- [Result] Korsatko S, Deller S, Koehler G, Mader JK, Neubauer K, Adrian CL, Thomsen H, Haahr H, Pieber TR. A comparison of the steady-state pharmacokinetic and pharmacodynamic profiles of 100 and 200 U/mL formulations of ultra-long-acting insulin degludec. Clin Drug Investig. 2013 Jul;33(7):515-21. doi: 10.1007/s40261-013-0096-7. PMID 23749405
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com